CLINICAL TRIAL: NCT05708963
Title: Occupational Physical Health Issues, Stress, Fatigue, and Burnout Experienced by U.K. Embryologists
Brief Title: The U.K. Embryologist Fatigue Study
Acronym: FUSE-UK
Status: Completed | Type: Observational
Sponsor: TMRW Life Sciences (Industry)
Collaborators: Dudley Associates Healthcare Marketing & Communications (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00062375-2
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Fatigue; Stress; Burnout, Professional; Musculoskeletal Pain; Back Pain; Neck Pain; Headache; Dizziness; Sleep Disturbance; Chest Pain; Syncope; Cardiovascular Diseases; Shortness of Breath; Gastrointestinal Diseases
Keywords: fatigue; burnout; stress; occupational health; occupational challenges
MeSH Terms: conditions — Fatigue; Burnout, Professional; Musculoskeletal Pain; Back Pain; Neck Pain; Headache; Dizziness; Parasomnias; Chest Pain; Syncope; Cardiovascular Diseases; Dyspnea; Gastrointestinal Diseases; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- U.K. Embryologists: U.K. embryologists of all ages, career levels, and other sociodemographic groups will be asked questions about their physical and mental health related to their occupational characteristics using the nationally validated surveys and questionnaires, and also about their working conditions in the ART/IVF laboratories using a custom occupational questionnaire and the single-item work unit grade (A-F).

SUMMARY:
The purpose of the study is to determine physical and mental health issues of U.K. embryologists related to their occupational characteristics, and how workplace fatigue and burnout may affect their quality of life, cynicism, interactions with patients, attention to detail, and lead to human error, the cause of the most severe IVF incidents that often make headlines and result in costly litigation. It will also correlate how the current manual workflows contribute to these health issues, and what measures can be taken to improve both working conditions and embryologists' health, and, therefore, improve patient care.

DETAILED DESCRIPTION:
Embryologist fatigue surveys conducted in Spain, the United States, and the international survey of embryologists from 85 countries reported that embryologists experience work-related fatigue, stress, and burnout. They named those as contributing factors to decreased efficiency, cynicism, and emotional exhaustion, which, together with having to handle the increasing cycle volume using conventional, manual protocols of cryomanagement, can lead to human error and IVF incidents. The known IVF incidents resulted in lost, damaged, or misplaced embryos and gametes, lawsuits, and reputational damage to patients and providers. In the absence of a "better than" cryopreservation storage solution, many programs just turned to buying more tanks and alarms and/or added expensive staff. The more effective solutions should focus on optimizing workflows by adopting innovation like automation and a digital chain of custody, organizational changes that will lead to a more productive, collaborative, and rewarding work environment, allowing embryologists to focus on patient care, scientific research, innovation, and career planning, and fewer incidents and lawsuits.

The purpose of this cross-sectional study using a web-based survey is to determine physical and mental health issues of U.K. embryologists related to their occupational characteristics, and how workplace fatigue and burnout may affect their quality of life, cynicism, interactions with patients, attention to detail, and lead to human error, the cause of the most severe IVF incidents that often make headlines and result in costly litigation. It will also correlate how the current manual workflows contribute to these health issues, and what measures can be taken to improve both working conditions and embryologists' health, and, therefore, improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* complete surveys from embryologists

Exclusion Criteria:

* incomplete surveys from embryologists; complete and incomplete surveys from non-embryologists.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Embryologists are the ART/IVF/embryology laboratory personnel who provide fertility and embryology services, including but not limited to IVF procedures, pre-implantation genetic testing of embryos, freezing/vitrification of embryos and gametes, cryomanagement of frozen/vitrified embryos and gametes, and monitoring and maintenance of laboratory records and equipment. They range in age, gender, marital status, children, and relationship status, but they must have a minimum of BA/BS degree, and HFEA or other professional certifications to work as an HFEA-licensed embryology laboratory technologist or supervisor, and a postgraduate degree, such as MA/MSci, PhD, MD, or DO to serve as the embryology laboratory director. Embryologists of all career levels work in a private, academic, government, or corporate IVF clinical/laboratory on a full-time, part-time, or per-diem basis, and with a permanent or a non-permanent contract.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
The sociodemographic characteristics of U.K. embryologists | 4-6 weeks
  The sociodemographic characteristics of U.K. embryologists whose routine work duties include IVF procedures and freezing and cryomanagement of embryos and gametes.
The work-related health status of U.K. embryologists | 4-6 weeks
  The overall health status of U.K. embryologists and associated health issues related to their professional duties.
The work-related stress and fatigue among U.K. embryologists | 4-6 weeks
  The stress and fatigue experienced by U.K. embryologists because of their reliance on manual procedures, the need for a high degree of attention to avoid errors and litigation and depending on human intervention to respond to emergencies in the laboratory.
The work-related burnout amount U.K. embryologists | 4-6 weeks
  The burnout experienced by U.K. embryologists because of their stress and fatigue.
Potential strategies to reduce stress, fatigue, and burnout in U.K. Embryologists | 4-6 weeks
  The potential strategies, such as organizational changes and automation of cryomanagement protocols, to alleviate physical strain and stress, and to prevent fatigue and burnout that can reduce the embryologist's attention to detail and contribute to IVF errors.

SECONDARY OUTCOMES:
The underlying causes of work-related physical and mental health issues in U.K. Embryologists | 4-6 weeks
  The underlying causes of physical strain, stress, fatigue, and burnout in U.K. embryologists related to their occupational characteristics.
The correlation between negative health outcomes, manual workload, and error among U.K. embryologists | 4-6 weeks
  How we can correlate these negative health outcomes and potential for human error they can cause, and link them to the overreliance of embryologists on outdated technology that adds time and stress to their workload.

CONTACTS AND LOCATIONS:
Overall Officials: Anar Murphy, PhD, Principal Investigator — TMRW Life Sciences
Locations (1):
- TMRW Life Sciences, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
TMRW and Dudley Associates (DA) will keep a master list containing personal identifiers and responses separate from data forms (paper and electronic) that have only analyzed results. The master list will be on a separate computer at DA. This form of data is considered "coded" not de-identified. Since the data can be re-linked to identifiers, it is coded. Only after the key to the code or the Master List is destroyed are the data considered de-identified. External investigators will not have access to these files
  The password-protected data will be stored on TMRW's drives in addition to the PIs' computers that are backed up according to TMRW's company policies
  The coded data with personally identifiable information of the survey participants will be stored as described above. The participants' personal identifiers and other data will be destroyed, and data will hence be de-identified 5 years after study completion in compliance with TMRW Data Classification and Handling Policy
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The coded preliminary data will become available on January 26, 2022, and it will be available to other researchers at TMRW and external collaborators for a limited duration of time, while preparing the abstract for the conference, and writing and revising a paper for a peer-reviewed publication. Only TMRW Principal Investigators and Dudley Associates will have access to the master file and participants' personal identifiers for 5 years. The participants' personal identifiers and other data will be destroyed, and data will, therefore, be de-identified 5 years after study completion in compliance with TMRW Data Classification and Handling Policy.
Access Criteria: All data and records generated during this survey will be kept confidential according to TMRW and Dudley Associates' policies on subject privacy and that the PIs and other TMRW personnel will not use them for any purpose other than conducting the study.
  All data will be anonymized by DA, and no record with personal identifiers will be available to anyone except for DA and TMRW PIs. TMRW's collaborators will be bound by the NDA, protecting the data and scientific integrity of this study.
  External collaborators will only be responsible for the data analysis, interpretation of the results, and co-authoring the abstract and a full peer-reviewed article using the coded data.
  No identifiable data will be used for future study without first obtaining REC approval or REC determination of exemption. The investigator will obtain a data use agreement between the provider (TMRW PIs) and any recipient researchers before sharing a limited dataset.

REFERENCES:
- [Background] Lopez-Leria B, Jimena P, Clavero A, Gonzalvo MC, Carrillo S, Serrano M, Lopez-Regalado ML, Olvera C, Martinez L, Castilla JA. Embryologists' health: a nationwide online questionnaire. J Assist Reprod Genet. 2014 Dec;31(12):1587-97. doi: 10.1007/s10815-014-0352-7. Epub 2014 Oct 5. PMID 25284212
- [Background] Tawfik DS, Profit J, Morgenthaler TI, Satele DV, Sinsky CA, Dyrbye LN, Tutty MA, West CP, Shanafelt TD. Physician Burnout, Well-being, and Work Unit Safety Grades in Relationship to Reported Medical Errors. Mayo Clin Proc. 2018 Nov;93(11):1571-1580. doi: 10.1016/j.mayocp.2018.05.014. Epub 2018 Jul 9. PMID 30001832
- [Background] Priddle H, Pickup S, Hayes C; Association of Reproductive and Clinical Scientists (ARCS). Occupational health issues experienced by UK embryologists: informing improvements in clinical reproductive science practice. Hum Fertil (Camb). 2022 Oct;25(4):608-617. doi: 10.1080/14647273.2021.1871782. Epub 2021 Jan 18. PMID 33459106
- [Background] West CP, Dyrbye LN, Shanafelt TD. Physician burnout: contributors, consequences and solutions. J Intern Med. 2018 Jun;283(6):516-529. doi: 10.1111/joim.12752. Epub 2018 Mar 24. PMID 29505159
- [Background] Frone MR, Tidwell MO. The meaning and measurement of work fatigue: Development and evaluation of the Three-Dimensional Work Fatigue Inventory (3D-WFI). J Occup Health Psychol. 2015 Jul;20(3):273-288. doi: 10.1037/a0038700. Epub 2015 Jan 19. PMID 25602275
- [Background] Shanafelt TD, West CP, Sinsky C, Trockel M, Tutty M, Satele DV, Carlasare LE, Dyrbye LN. Changes in Burnout and Satisfaction With Work-Life Integration in Physicians and the General US Working Population Between 2011 and 2017. Mayo Clin Proc. 2019 Sep;94(9):1681-1694. doi: 10.1016/j.mayocp.2018.10.023. Epub 2019 Feb 22. PMID 30803733
- [Background] Trockel MT, Menon NK, Rowe SG, Stewart MT, Smith R, Lu M, Kim PK, Quinn MA, Lawrence E, Marchalik D, Farley H, Normand P, Felder M, Dudley JC, Shanafelt TD. Assessment of Physician Sleep and Wellness, Burnout, and Clinically Significant Medical Errors. JAMA Netw Open. 2020 Dec 1;3(12):e2028111. doi: 10.1001/jamanetworkopen.2020.28111. PMID 33284339
- [Background] Caruso CC, Baldwin CM, Berger A, Chasens ER, Edmonson JC, Gobel BH, Landis CA, Patrician PA, Redeker NS, Scott LD, Todero C, Trinkoff A, Tucker S. Policy brief: Nurse fatigue, sleep, and health, and ensuring patient and public safety. Nurs Outlook. 2019 Sep-Oct;67(5):615-619. doi: 10.1016/j.outlook.2019.08.004. No abstract available. PMID 31582105
- [Background] Dyrbye LN, Shanafelt TD, Johnson PO, Johnson LA, Satele D, West CP. A cross-sectional study exploring the relationship between burnout, absenteeism, and job performance among American nurses. BMC Nurs. 2019 Nov 21;18:57. doi: 10.1186/s12912-019-0382-7. eCollection 2019. PMID 31768129
- [Background] Letterie G, Fox D. Lawsuit frequency and claims basis over lost, damaged, and destroyed frozen embryos over a 10-year period. F S Rep. 2020 Jul 9;1(2):78-82. doi: 10.1016/j.xfre.2020.06.007. eCollection 2020 Sep. PMID 34223222
- [Background] Moutos CP, Lahham R, Phelps JY. Cryostorage failures: a medicolegal review. J Assist Reprod Genet. 2019 Jun;36(6):1041-1048. doi: 10.1007/s10815-019-01478-x. Epub 2019 May 24. PMID 31127476
- [Background] Boivin J, Bunting L, Koert E, Ieng U C, Verhaak C. Perceived challenges of working in a fertility clinic: a qualitative analysis of work stressors and difficulties working with patients. Hum Reprod. 2017 Feb;32(2):403-408. doi: 10.1093/humrep/dew326. Epub 2017 Jan 5. PMID 28057875
- [Background] Applebaum J, Humphries LA, Nepps ME, Berger DS, O'Neill K. Malpractice litigation surrounding in vitro fertilization in the United States: a legal literature review. Fertil Steril. 2023 Apr;119(4):572-580. doi: 10.1016/j.fertnstert.2022.12.038. Epub 2022 Dec 27. PMID 36581015
- [Derived] Murphy A, Lapczynski MS, Proctor G Jr, Glynn TR, Domar AD, Gameiro S, Palmer GA, Collins MG. Comparison of embryologist stress, somatization, and burnout reported by embryologists working in UK HFEA-licensed ART/IVF clinics and USA ART/IVF clinics. Hum Reprod. 2024 Oct 1;39(10):2297-2304. doi: 10.1093/humrep/deae191. PMID 39198005
- See also: The Human Fertilisation & Embryology Authority. Fertility treatment 2019: trends and figures. UK statistics for IVF and DI treatment, storage, and donation. May 2021. — https://www.hfea.gov.uk/about-us/publications/research-and-data/fertility-treatment-2019-trends-and-figures/
- See also: The Human Fertilisation & Embryology Authority. How we regulate — https://www.hfea.gov.uk/about-us/how-we-regulate/
- See also: The Human Fertilisation & Embryology Authority. The Code of practice. 9th Edition. 2021. — https://www.hfea.gov.uk/about-us/news-and-press-releases/2021-news-and-press-releases/update-to-the-9th-edition-code-of-practice-is-now-available/
- See also: The Human Fertilisation & Embryology Authority. State of the fertility sector 2019/2020. November 2020. — https://www.hfea.gov.uk/about-us/publications/research-and-data/state-of-the-fertility-sector-2019-2020/
- See also: Embryologist burnout: physical and psychological symptoms and occupational challenges currently reported by U.S. embryologists — https://doi.org/10.1016/j.fertnstert.2022.08.205
- See also: Working with fatigue: assessment of cryomanagement conditions in IVF biorepositories — https://doi.org/10.1016/j.fertnstert.2022.08.368
- See also: A Pragmatic Approach for Organizations to Measure Health Care Professional Well-Being — https://nam.edu/a-pragmatic-approach-for-organizations-to-measure-health-care-professional-well-being/